CLINICAL TRIAL: NCT02483039
Title: Nephrologist Follow-up Versus Usual Care After an Acute Kidney Injury Hospitalization (FUSION): Vanguard Phase of a Randomized Controlled Trial
Brief Title: Nephrologist Follow-up Versus Usual Care After an Acute Kidney Injury Hospitalization
Acronym: FUSION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Unity Health Toronto (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other); University Health Network, Toronto (Other); Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 004
Record Dates: First submitted 2015-06-18; First posted 2015-06-26 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Acute Kidney Injury; Chronic Kidney Disease
Keywords: Acute kidney injury; Chronic kidney disease; Quality improvement
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AKI Follow-up Clinic (Experimental): Participants randomized to this arm will be referred to the AKI Follow-up Clinic where they will see a nephrologist who will coordinate follow-up care. The target appointment date is within 30 days of hospital discharge. Routine laboratory investigations will be performed at minimum every three months. Additional in-person visits with a nephrologist at the AKI Follow-up Clinic will be determined at the local sites based upon the participant's clinical status. If in-person visits at 12, 24, and/or 36 weeks are not necessary given the patient's clinical status, they may be replaced with a telephone visit
  Interventions: Behavioral: AKI Follow-up Clinic
- Usual Care (No Intervention): Participants randomized to this arm will have a letter outlining their AKI diagnosis mailed to their family physician. Participants may still be referred to a nephrologist by their inpatient or outpatient healthcare provider, but these participants will not have access to the AKI Follow-up Clinic. Rather, they will proceed through the standard local nephrology referral pathway. In addition, all usual care participants will be contacted via telephone by study staff every three months to assess their clinical condition and ensure study engagement. All usual care participants will be offered a nephrologist assessment and/or bloodwork one year after randomization to determine if ongoing nephrology care is indicated based upon the same criteria applied to AKI Follow-up Clinic participants.

INTERVENTIONS:
Behavioral: AKI Follow-up Clinic — Participants randomized to this arm will be referred to the AKI Follow-up Clinic where they will see a nephrologist who will coordinate follow-up care. At the AKI Follow-up Clinic, assessment forms that were developed during the pilot study at St. Michael's Hospital may be used, but this decision will be left to individual sites. Routine laboratory investigations will be performed at minimum every three months.
  Arms: AKI Follow-up Clinic

SUMMARY:
The primary objective is to evaluate the impact of an AKI Follow-up Clinic on major adverse kidney events (MAKE) in comparison to hospitalized patients surviving an episode of AKI who are not exposed to the AKI Follow-up Clinic intervention.

DETAILED DESCRIPTION:
Survivors of acute kidney injury (AKI) are at increased risk of chronic kidney disease (CKD) and death, but have inconsistent follow-up care. Our team has developed and tested a model to deliver structured follow-up kidney care (the AKI Follow-up Clinic) that is feasible and sustainable, with standardized assessments based upon clinical practice guidelines that are transferable to any setting. This study will randomize patients with Kidney Disease Improving Global Outcomes (KDIGO) stage 2-3 AKI to the AKI Follow-up Clinic or usual care (control group). The usual care group will have a letter outlining their AKI diagnosis mailed to their family physician; the usual care group may still be referred to a nephrologist by their healthcare provider if desired, but these participants will not have access to the AKI Follow-up Clinic pathways. The primary outcome is development of a major adverse kidney event (MAKE), a composite of death, chronic dialysis, and estimated glomerular filtration rate (eGFR) decline. Outcomes will be ascertained after one year of follow-up, which is when AKI Follow-up Clinic patients are transitioned back to their family doctor or general nephrologist based upon pre-specified graduation criteria. Participants will also be followed using local hospital electronic resources and the Institute for Clinical Evaluative Sciences (ICES) administrative databases in order to assess the long-term impact of early nephrologist follow-up on AKI outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 yrs
* Kidney Disease Improving Global Outcomes (KDIGO) stage 2 AKI and above (including need for dialysis)

Exclusion Criteria:

* Kidney transplant recipients
* Outpatient baseline eGFR under 30mL/min/1.73m2 (by CKD-EPI equation); ignore if baseline serum creatinine is unavailable
* Patients discharged from hospital with a persistent requirement for renal replacement therapy
* Clinical diagnosis or suspicion of: glomerulonephritis, vasculitis with kidney involvement, hemolytic-uremic syndrome, polycystic kidney disease, myeloma cast nephropathy
* Pregnancy
* Residence at a nursing home facility (rehabilitation and retirement home patients should not be excluded)
* Palliation as primary goal of care (defined as life expectancy ≤ six months or followed by a palliative care physician)
* Patients with previously established and ongoing nephrology follow-up (defined as ≥ one outpatient appointment with a nephrologist in the previous 12 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-09; Primary Completion 2018-07 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Proportion with a major adverse kidney event | 1 year after randomization
  Composite of chronic dialysis, chronic kidney disease progression, or death

SECONDARY OUTCOMES:
Proportion with a major adverse kidney event | 30, 90, 365 days, and 5 years following randomization
  Composite of chronic dialysis, chronic kidney disease progression, or death
Proportion deceased | 30, 90, 365 days, and 5 years following randomization
Proportion who require chronic dialysis | 30, 90, 365 days, and 5 years following randomization
  one outpatient dialysis treatment at any time after randomization
Proportion with chronic kidney disease progression using CKD-EPI eGFR equation | 30, 90, 365 days, and 5 years following randomization
Time to major adverse kidney event | 5 years following randomization
  Composite of chronic dialysis, chronic kidney disease progression, or death
Time to death | 5 years following randomization
Time to chronic dialysis | 5 years following randomization
  one outpatient dialysis treatment at any time after randomization
Time to CKD progression using CKD-EPI eGFR equation | 5 years following randomization
Proportion with a major adverse cardiac event | 30, 90, 365 days, and 5 years following randomization
  Defined as a hospitalization or emergency department visit for stroke, congestive heart failure, myocardial infarction, or cardiac revascularization procedure
Proportion who experience a stroke | 30, 90, 365 days, and 5 years following randomization
  Hospitalization or emergency department visit for stroke
Proportion who experience a congestive heart failure episode | 30, 90, 365 days, and 5 years following randomization
  Hospitalization or emergency department visit for congestive heart failure
Proportion who undergo a cardiac revascularization procedure | 30, 90, 365 days, and 5 years following randomization
  Hospitalization or emergency department visit for a cardiac revascularization procedure
Proportion who experience a myocardial infarction | 30, 90, 365 days, and 5 years following randomization
  Hospitalization or emergency department visit for myocardial infarction
Time to first rehospitalization | 5 years following randomization
  Defined as the first readmission to hospital for any reason
Time to first emergency department visit | 5 years post-randomization
  Defined as the first emergency department visit for any reason
Time to first acute kidney injury episode post-randomization using KDIGO serum creatinine criteria | 5 years post-randomization
Number of acute kidney injury episodes post-randomization using KDIGO serum creatinine criteria | 5 years post-randomization
Change in quality-of-life as measured by EuroQol-5D-5L instrument | 1 year post-randomization

CONTACTS AND LOCATIONS:
Overall Officials: Ron Wald, MDCM, MPH, Principal Investigator — Unity Health Toronto
Locations (4):
- Canada (4):
  - Mount Sinai Hospital, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario

REFERENCES:
- [Derived] Robinson C, Hessey E, Nunes S, Dorais M, Chanchlani R, Lacroix J, Jouvet P, Phan V, Zappitelli M. Acute kidney injury in the pediatric intensive care unit: outpatient follow-up. Pediatr Res. 2022 Jan;91(1):209-217. doi: 10.1038/s41390-021-01414-9. Epub 2021 Mar 17. PMID 33731806